CLINICAL TRIAL: NCT04659642
Title: Attenuation of Airway and Cardiovascular Responses to Extubation in Chronic Smokers by Prior Treatment With Dexmedetomidine, Fentanyl and Their Combination
Brief Title: Attenuation of Airway and Cardiovascular Responses to Extubation in Chronic Smokers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Asmaa Fahmy Mohamed Abdelwahab, Doctor, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: dexmedetomidine in anesthesia
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Airway Responses; Hemodynamic
Keywords: extubation; chronic smoker; dexmedetomidine; fentanyl; abdominal surgery
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- dexmedetomidine group (group A) (Active Comparator): will receive Dexmedetomidine 1ug/kg body weight IV diluted to 100ml normal saline (NS) over 15 minutes.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Fentanyl group (group B) (Active Comparator): will receive Fentanyl 1 ug/kg body weight IV diluted to 100 ml normal saline (NS) over 15 minutes.
  Interventions: Drug: Fentanyl Citrate Injection
- Both Dexmedetomidine and fentanyl group (group C) (Active Comparator): will receive both Dexmedetomidine 1ug/kg body weight mixed with fentanyl 1ug/kg in 100 ml normal saline (NS) over 15 minutes.
  Interventions: Combination Product: dexmedetomidine and fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — the drug is given 15 minutes before the estimated end of surgery
  Arms: dexmedetomidine group (group A)
Drug: Fentanyl Citrate Injection — the drug is given 15 minutes before the estimated end of surgery
  Arms: Fentanyl group (group B)
Combination Product: dexmedetomidine and fentanyl — the combination of the two drugs with the same used doses is given 15 minutes before the estimated end of surgery
  Arms: Both Dexmedetomidine and fentanyl group (group C)

SUMMARY:
The aim of this blind comparative study was to compare the effects of dexmedetomidine, fentanyl and their combination on airway reflexes and hemodynamic responses to tracheal extubation in Adult chronic male smoking patients scheduled for abdominal surgeries (of average 2-3 hours duration).

DETAILED DESCRIPTION:
Tracheal extubation is associated with acute, transient, significant and undesirable hemodynamic and airway responses that may persist into the recovery period. Respiratory complications after tracheal extubation are three times more common than complications occurring during tracheal intubation and induction of anesthesia (4.6% vs 12.6%) .

The peak changes are noticed about 1 minute following extubation and may continue until 10 minutes . The reflexes ranges from coughing, bucking, agitation to bronchospasm, laryngospasm, laryngeal oedema, negative pressure pulmonary oedema, tachycardia, hypertension, arrhythmias, left ventricular failure, myocardial ischemia, increased bleeding, raised intracranial and intraocular pressure and cerebrovascular hemorrhage in susceptible individuals. Although most patients can tolerate these transient effects without any significant consequences, but this could be detrimental in patients operated for cardiac, neuro or ophthalmic lesions especially if hypertensive or diabetic. However, Tracheal extubation in smokers will increase difficulty.

Smoking is a risk factor for intraoperative and postoperative complications mainly related to pulmonary and cardiovascular systems. Long-term exposure to cigarettes causes an increased response to the mechanical stimulation caused by extubation.

Smoking affects oxygen transport and delivery , Irritants in smoke increase mucous secretion which becomes hyper viscous with impaired tracheobronchial clearance . Smoking increases sympathetic activation due to increased release of catecholamines and the delay in nicotine clearance from the neuroeffector junction leading to higher blood pressure, tachycardia, and increase peripheral vascular resistance .

For a smooth extubation, there should be no straining, movement, coughing, breath holding or laryngospasm. Extubation at light levels of anesthesia or sedation can stimulate reflex responses via tracheal and laryngeal irritation . A variety of drugs such as esmolol, alfentanil, diltiazem, verapamil, fentanyl, and lidocaine have been used to control hemodynamic changes and upper airway tract events, but they all have limitations and side effects.

Alpha2 agonists decrease the sympathetic outflow and noradrenergic activity, thereby counteracting hemodynamic fluctuations occurring at the time of extubation due to increased sympathetic stimulation. Dexmedetomidine, an α2-adrenoreceptor agonist with a distribution half-life of approximately 6 minutes has been successfully used for attenuating the stress response to laryngoscopy .

Single dose of dexmedetomidine before extubation proved to attenuate both airway and hemodynamic reflexes during emergence from anesthesia providing smooth extubation.

The addition of a single dose of dexmedetomidine to a low-dose infusion of remifentanil during emergence from sevoflurane-remifentanil anesthesia was effective in attenuating cough without further respiratory depression after thyroid surgery.

Administered 10 minutes before induction in chronic male smokers, dexmedetomidine was found to suppress increased heart rate and rate-pressure product at 1 and 3 minutes after intubation and, therefore, decrease the need for myocardial oxygen more than fentanyl.

Dexmedetomidine produces sedation while sparing responsiveness to CO2, and thus, it has less effect on respiratory depression. Consequently, it has found utility and regulatory approval for use in bronchoscopic examinations and for weaning intensive care unit patients from mechanical ventilation. In addition, dexmedetomidine has been shown to reduce emergence agitation in children and adults after general anesthesia.

Fentanyl, a synthetic opioid, has been reported to reduce the prevalence of coughing during and after extubation and to suppress the sneezing reflex after abdominal hysterectomy and periocular injections . Fentanyl has also been reported to attenuate the cardiovascular responses to tracheal extubation in elective gynecologic surgery.

The subjects were Adult chronic male smokers, thus representing the population in which secondary response to laryngoscopy and intubation is most common.

The study participants will be divided by mean of randomized complete block design into 3 comparable groups.

Group (A) : (n= 22) will receive Dexmedetomidine 1ug/kg body weight IV diluted to 100ml normal saline (NS) over 15 minutes.

Group (B) : (n=22) will receive Fentanyl 1 ug/kg body weight IV diluted to 100 ml normal saline (NS) over 15 minutes.

Group (C): (n=22) will receive both Dexmedetomidine 1ug/kg body weight mixed with fentanyl 1ug/kg in 100 ml normal saline (NS) over 15 minutes Pre-anesthetic checkup was conducted and a detailed history and complete physical examination recorded. Routine investigations like complete blood picture, blood grouping/typing, blood urea and serum creatinine were done. Patients fulfilling inclusion criteria will be informed about the procedure and its possible complications. Finally, written consent will be taken.

Routine anesthetic technique was used using propofol 2mg/kg, fentanyl 1.5 ug/kg, atracurium 0.5 mg /kg, oxygen and sevoflurane. Standard monitoring with electrocardiography (EKG), pulse oximetry (SpO2), noninvasive BP and End tidal Co2 was done.

About 15 minutes before the estimated time of end of surgery (or at the beginning of closure of skin incision,), inhalation agent (sevoflurane) was cut off and patients in each group received the specified solution intravenously over 15 minutes.

Patients in group A received dexmedetomidine 1 mcg/kg intravenous (IV) in 100 ml normal saline (NS) over 15 minutes ,patients in group B, received Fentanyl 1 mcg/kg (IV) in100 ml NS over 15 minutes, while patients in group C received both Dexmedetomidine 1ug/kg mixed with fentanyl 1ug/kg in 100 ml normal saline (NS) over 15 minutes.

When patients' spontaneous respirations were considered sufficient and patients were able to obey simple commands residual neuromuscular block was antagonized with neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Oropharyngeal secretions were aspirated before extubation. The endotracheal tube was removed after spontaneous ventilation had returned.

The anesthesiologist performing the extubation was blinded to the study drugs. HR, systolic BP and diastolic BP and oxygen saturation were recorded at the start of bolus drug injection and thereafter at 1, 3, 5, 10 and 15 minutes., Also at the time of extubation and thereafter at 1, 3 and 5 minutes after extubation followed by every 5 minutes for 30 minutes. Duration of anesthesia and surgery are noted.

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 22 (SPSS Inc., Chicago, IL). Numerical data will be described as median and interquartile range or range or mean and standard deviation as appropriate, while qualitative data were described as number and percentage. Chi-square (Fisher's exact) test was used to examine the relation between qualitative variables as appropriate. Testing for normality was done using Kolmogrov-Smirnov test and Shapiro-Wilk test

ELIGIBILITY:
Inclusion Criteria:

* Chronic cigarette smokers (patients have smoked for two years at least, and a minimum consumption of 10 cigarettes/ day)
* American Society of Anesthesiologists (ASA) II.
* Normotensive and receiving no medications
* Body mass index of 30 kg/m2
* Mallampati classification I-II

Exclusion Criteria:

1. History of opioid, sedative drugs or medications affecting heart rate or blood pressure.
2. Morbid obesity.
3. Current upper respiratory infection
4. Hypovolemia
5. IHD
6. History of sleep apnea or Difficult Intubation.
7. Emergency procedures.
8. Hepatic or renal impairment.
9. Drug allergy to Dexmeditomidine or fentanyl.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-03-06 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
Quality of extubation by extubation quality score | 5 minutes
  1. No coughing
  2. Smooth extubation, minimal coughing (1 or 2 times)
  3. Moderate coughing (3 or 4 times)
  4. Severe coughing (5-10 times) and straining
  5. Poor extubation, very uncomfortable (laryngospasm and coughing >10 times).
post extubation laryngospasm, bronchospasm or desaturation | 30 minutes
  laryngospasm, bronchospasm or desaturation

SECONDARY OUTCOMES:
Time to extubation | up to 25 minutes
  from inhaled anesthetic cut off to ETT removal
Hemodynamic responses | up to 60 minutes
  Bradycardia (was defined as HR < 60 /min and treated with rescue dose of injection atropine 0.6 mg intravenously), tachycardia (being 20% increase from baseline), hypertension (as either 20% increase from baseline or SBP > 180 mmHg) and hypotension (as 20% decrease from baseline or SBP < 80 mmHg).
• Postoperative agitation and sedation were evaluated on a 10 points scale (RASS Scale) | up to 30 minutes
  (+4) Combative, (+3) Very Agitated, (+2) Agitated, (+1) Restless, (0) Alert and Calm, (-1) Drowsy, (-2) Light sedation, (-3) Moderate sedation, (-4) Deep sedation, (-5) Unarousable.

CONTACTS AND LOCATIONS:
Overall Officials: naglaa abdullah, prof, Principal Investigator — NCI, Cairo university
Locations (1):
- NCI, Cairo university, Cairo, Egypt